CLINICAL TRIAL: NCT01210482
Title: SAFETY AND EFFECTIVENESS OF TEMSIROLIMUS IN JAPANESE PATIENTS WITH UNRESECTABLE OR METASTATIC RENAL CELL CARCINOMA: A POST-MARKETING, ALL-CASE SURVEILLANCE STUDY INCLUDING B1771016 STUDY - SURVEY ON LONG-TERM USE -
Brief Title: Temsirolimus (Torisel) Drug Use Investigation (Regulatory Post Marketing Commitment Plan)
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 3066K5-4406; B1771015 (Other: Alias Study Number); NCT01420601 (obsolete NCT alias)
Record Dates: First submitted 2010-09-27; First posted 2010-09-28 (Estimated); Results first posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-06

CONDITIONS: Renal Cell Carcinoma
Keywords: Torisel; Regulatory Post Marketing Commitment Plan
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — temsirolimus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Temsirolimus: Patients treated with Torisel (patients with metastatic and/or radically unresectable or advanced renal cell carcinoma)
  Interventions: Drug: Temsirolimus

INTERVENTIONS:
Drug: Temsirolimus — The usual adult dosage is temsirolimus 25 mg once weekly, to be administered via gradual intravenous infusion over 30~60 minutes. The dosage is to be appropriately reduced according to patients' status.
  Other Names: Torisel

SUMMARY:
The objective of this investigation is to determine the following items in all patients receiving Torisel for a certain period after marketing:

1. Confirmation of efficacy and safety for medical practice use.
2. Investigation of factors that may influence the incidence of adverse events (Particularly priority investigation items).
3. Investigation of the incidence status and the risk factors for interstitial lung diseases.

DETAILED DESCRIPTION:
Implemented as a Drug Use Investigation by Central Registration System

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with Torisel (patients with metastatic and/or radically unresectable or advanced renal cell carcinoma).

Exclusion Criteria:

* Patients not administered Torisel.
* Patients with a history of severe hypersensitivity to temsirolimus, sirolimus derivative, or any of their components and/or derivatives.

Ages: 15 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated with Torisel (patients with metastatic and/or radically unresectable or advanced renal cell carcinoma).
Sampling Method: Probability Sample
Enrollment: 1050 (Actual)
Dates: Start 2010-08-24 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Kyusyu University Hospital, Fukuoka, Fukuoka PREF, Japan

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Sugiyama S, Sato K, Shibasaki Y, Endo Y, Uryu T, Toyoshima Y, Oya M, Miyanaga N, Saijo N, Gemma A, Akaza H. Real-world use of temsirolimus in Japanese patients with unresectable or metastatic renal cell carcinoma: recent consideration based on the results of a post-marketing, all-case surveillance study. Jpn J Clin Oncol. 2020 Aug 4;50(8):940-947. doi: 10.1093/jjco/hyaa062. PMID 32458996
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3066K5-4406&StudyName=Temsirolimus%20%28Torisel%29%20Drug%20Use%20Investigation%20%28Regulatory%20Post%20Marketing%20Commitment%20Plan%29

RESULTS

PARTICIPANT FLOW:
Groups:
- TORISEL Injection (Temsirolimus): Patients prescribed temsirolimus for its approved indication (radically unresectable or metastatic RCC) were registered and received temsirolimus in routine clinical settings (observation period: 96 weeks)
Period: Overall Study
Arm/Group | TORISEL Injection (Temsirolimus)
Started | 1050
Completed | 1001
Not Completed | 49
Not completed — Protocol Violation | 1
Not completed — Case Report Forms were not collected | 18
Not completed — Duplicated | 2
Not completed — No Drug Administration | 28

BASELINE CHARACTERISTICS:
Population: A total of 1050 participants were enrolled in this study. Of the 1050 participants, 49 participants were excluded from the safety analysis set due to following reasons: no drug administration (28 participants), duplication (2 participants), case report forms were not collected (18 participants), protocol violation (1 participant).
Arm/Group | TORISEL Injection (Temsirolimus)
Number analyzed (Participants) | 1001
Age, Customized [Number; unit: Participants]
  < 15 years | 3
  ≥ 15 and < 65 years | 489
  ≥ 65 years | 493
  Unknown | 16
Sex/Gender, Customized [Number; unit: Participants]
  Male | 749
  Female | 252
Race/Ethnicity, Customized [Number; unit: Participants]
  Race and Ethnicity Not Collected | 1001

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Drug Reactions
Description: An adverse drug reaction (ADR) was any untoward medical occurrence attributed to TORISEL Injection in a participant who received TORISEL Injection. A serious ADR was an ADR resulting in any of the following outcomes or deemed significant for any other reason: death, life-threatening experience (immediate risk of dying), initial or prolonged inpatient hospitalization, persistent or significant disability/incapacity, congenital anomaly. Relatedness to TORISEL Injection was assessed by the physician.
Time Frame: 96 weeks at maximum
Population: The safety analysis set comprised of participants who satisfied the inclusion criteria and had received TORISEL Injection at least once.
Measure: Number; unit: Participants
Arm/Group | TORISEL Injection (Temsirolimus)
Number analyzed (Participants) | 1001
Participants
  ADR | 778
  Serious ADR | 352

2. Primary Outcome: Number of Participants With Adverse Drug Reactions of Major Investigation Items
Description: An adverse drug reaction (ADR) was any untoward medical occurrence attributed to TORISEL Injection in a participant who received TORISEL Injection. Sixteen events were evaluated as major investigation items, and the result is presented in the table.
Time Frame: 96 weeks at maximum
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | TORISEL Injection (Temsirolimus)
Number analyzed (Participants) | 1001
Participants
  Mucositis related adverse events | 279
  Skin disorder | 209
  Interstitial lung disease | 174
  Interstitial lung disease suspected events | 3
  Infections | 141
  Hypercholesterolaemia/hyperlipidaemia | 140
  Diabetes/hyperglycaemia | 131
  Diarrhoea | 43
  Hypophosphataemia | 39
  Dyspnea | 35
  Acute renal failure | 17
  Hypokalaemia | 14
  Hypersensitivity reaction | 11
  Gastrointestinal perforation | 1
  Intracerebral hemorrhage | 1
  Wound healing abnormal | 1

3. Secondary Outcome: Overall Response Rate
Description: Clinical response was assessed based on the following 4 classes with reference to the "New response evaluation criteria in solid tumours: Revised RECIST guideline (version 1.1) - Japanese Translation JCOG Version:" complete response (CR), partial response (PR), progressive disease (PD), stable disease (SD). The overall response rate, which was defined as the percentage of participants who achieved CR or PR over the total number of assessable effectiveness analysis population, was presented along with the corresponding 2-sided 95% confidence interval.
Time Frame: 96 weeks maximum
Population: The efficacy analysis set is comprised in the safety analysis set who was considered to have undergone an appropriate evaluation.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | TORISEL Injection (Temsirolimus)
Number analyzed (Participants) | 654
Percentage of Participants | 6.7 [4.9 to 8.9]

4. Secondary Outcome: Response Rate Excluding Participants Evaluated as "Unassessable"
Description: Clinical response was assessed based on the following 4 classes with reference to the "New response evaluation criteria in solid tumours: Revised RECIST guideline (version 1.1) - Japanese Translation JCOG Version:" complete response (CR), partial response (PR), progressive disease (PD), stable disease (SD). The percentage of participants who achieved CR or PR over the total number of assessable effectiveness analysis population excluding those evaluated as "unassessable," was calculated.
Time Frame: 96 weeks maximum
Population: The efficacy analysis set is comprised in the safety analysis set who was considered to have undergone an appropriate evaluation (n=654). Of these, 63 participants were evaluated as "unassessable" in the analysis of clinical response.
Measure: Number; unit: Percentage of Participants
Arm/Group | TORISEL Injection (Temsirolimus)
Number analyzed (Participants) | 591
Percentage of Participants | 7.4

ADVERSE EVENTS:
Time Frame: 96 weeks maximum
Description: The frequency of adverse events. The same event may appear as both an adverse event and a serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both serious and non-serious events during the study.
Arm/Group | TORISEL Injection (Temsirolimus)
All-Cause Mortality (participants affected / at risk) | 185/1001
Serious Adverse Events (participants affected / at risk) | 499/1001
Other Adverse Events (participants affected / at risk) | 759/1001
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TORISEL Injection (Temsirolimus) (N=1001)
Shock (Vascular disorders) | 1
Flushing (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2
Drug eruption (Skin and subcutaneous tissue disorders) | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1
Sputum retention (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 15
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 174
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 40
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Renal impairment (Renal and urinary disorders) | 3
Renal failure (Renal and urinary disorders) | 3
Renal disorder (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Chronic kidney disease (Renal and urinary disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 12
Communication disorder (Psychiatric disorders) | 1
Seizure (Nervous system disorders) | 2
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1
Hemiplegia (Nervous system disorders) | 1
Embolic cerebral infarction (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 2
Cerebral haemorrhage (Nervous system disorders) | 1
Brain oedema (Nervous system disorders) | 1
Altered state of consciousness (Nervous system disorders) | 1
Akathisia (Nervous system disorders) | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 12
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 3
Decreased appetite (Metabolism and nutrition disorders) | 6
Cachexia (Metabolism and nutrition disorders) | 1
White blood cell count decreased (Investigations) | 7
Weight increased (Investigations) | 1
Protein urine (Investigations) | 1
Platelet count decreased (Investigations) | 10
Nutritional condition abnormal (Investigations) | 1
Neutrophil count decreased (Investigations) | 2
Lipase increased (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Glycosylated haemoglobin increased (Investigations) | 1
C-reactive protein increased (Investigations) | 1
Chest X-ray abnormal (Investigations) | 1
Blood uric acid increased (Investigations) | 1
Blood urea increased (Investigations) | 1
Blood pressure increased (Investigations) | 2
Blood glucose increased (Investigations) | 1
Blood creatinine increased (Investigations) | 5
Blood cholesterol increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Alanine aminotransferase increased (Investigations) | 1
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1
Injury (Injury, poisoning and procedural complications) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Wound infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Shunt infection (Infections and infestations) | 1
Septic shock (Infections and infestations) | 2
Sepsis (Infections and infestations) | 3
Respiratory tract infection (Infections and infestations) | 1
Rash pustular (Infections and infestations) | 1
Pseudomembranous colitis (Infections and infestations) | 1
Pneumonia staphylococcal (Infections and infestations) | 1
Pneumonia bacterial (Infections and infestations) | 15
Pneumonia (Infections and infestations) | 24
Pneumocystis jirovecii infection (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 3
Lung infection (Infections and infestations) | 2
Infection (Infections and infestations) | 3
Infected skin ulcer (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 4
Hepatitis B reactivation (Infections and infestations) | 1
Fungal infection (Infections and infestations) | 1
Cytomegalovirus enterocolitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 1
Atypical pneumonia (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 1
Anorectal infection (Infections and infestations) | 1
Anal abscess (Infections and infestations) | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 10
Immunosuppression (Immune system disorders) | 1
Hypersensitivity (Immune system disorders) | 2
Anaphylactic shock (Immune system disorders) | 2
Anaphylactic reaction (Immune system disorders) | 1
Liver disorder (Hepatobiliary disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 3
Cholecystitis (Hepatobiliary disorders) | 4
Biliary tract disorder (Hepatobiliary disorders) | 1
Sudden death (General disorders) | 1
Pyrexia (General disorders) | 6
Oedema (General disorders) | 5
Malaise (General disorders) | 2
Generalised oedema (General disorders) | 1
Gait disturbance (General disorders) | 1
Fatigue (General disorders) | 2
Disease progression (General disorders) | 145
Death (General disorders) | 5
Chest pain (General disorders) | 1
Asthenia (General disorders) | 1
Vomiting (Gastrointestinal disorders) | 5
Stomatitis (Gastrointestinal disorders) | 15
Pancreatitis acute (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 6
Large intestine perforation (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 3
Ileus paralytic (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 2
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Gastrointestinal perforation (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3
Enterocolitis (Gastrointestinal disorders) | 3
Dysphagia (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 5
Colitis ulcerative (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 2
Abdominal hernia (Gastrointestinal disorders) | 1
Visual impairment (Eye disorders) | 1
Diplopia (Eye disorders) | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Pericardial effusion (Cardiac disorders) | 2
Myocardial ischaemia (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 3
Cardiac failure acute (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 4
Cardiac arrest (Cardiac disorders) | 1
Atrioventricular block complete (Cardiac disorders) | 2
Acute myocardial infarction (Cardiac disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 4
Bone marrow failure (Blood and lymphatic system disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TORISEL Injection (Temsirolimus) (N=1001)
Stomatitis (Gastrointestinal disorders) | 257
Anaemia (Blood and lymphatic system disorders) | 59
Pyrexia (General disorders) | 54
Platelet count decreased (Investigations) | 104
Hypercholesterolaemia (Metabolism and nutrition disorders) | 56
Hyperglycaemia (Metabolism and nutrition disorders) | 93
Hyperlipidaemia (Metabolism and nutrition disorders) | 60
Rash (Skin and subcutaneous tissue disorders) | 76

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2011-02-02): https://cdn.clinicaltrials.gov/large-docs/82/NCT01210482/Prot_000.pdf
  • Statistical Analysis Plan (2016-09-26): https://cdn.clinicaltrials.gov/large-docs/82/NCT01210482/SAP_001.pdf